CLINICAL TRIAL: NCT06923800
Title: Comparison of Two Exercise Interventions and Dietary Advice in Patients With Fibromyalgia and Irritable Bowel Syndrome: A Randomized Controlled Crossover Study
Brief Title: Exercise Interventions and Dietary Advice in Fibromyalgia and IBS
Acronym: FM-IBS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Antonella Bianco, Principal Investigator, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AF_FM crossover
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Fibromyalgia; Irritable Bowel Syndrome
Keywords: exercise; aerobic exercise; fibromyalgia; irritable bowel syndrome
MeSH Terms: conditions — Fibromyalgia; Irritable Bowel Syndrome; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Masking Description: first treatment assignment is randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FM+IBS Group 1 (Experimental): Patients with Fibromyalgia and IBS
  Interventions: Behavioral: Combined Exercise Program + A specific nutritional plan for individuals with IBS; Behavioral: Aerobic Exercise + A specific nutritional plan for individuals with IBS
- FM + IBS Group 2 (Experimental): Patients with Fibromyalgia and IBS
  Interventions: Behavioral: Combined Exercise Program + A specific nutritional plan for individuals with IBS; Behavioral: Aerobic Exercise + A specific nutritional plan for individuals with IBS

INTERVENTIONS:
Behavioral: Combined Exercise Program + A specific nutritional plan for individuals with IBS — 60-minute sessions three times per week for 4 months, incorporating moderate aerobic, resistance, and flexibility exercises
Behavioral: Aerobic Exercise + A specific nutritional plan for individuals with IBS — 60-minute sessions, three times a week for 4 months, with low-impact, non-weight-bearing aerobic activities at 60-75% of max heart rate.

SUMMARY:
Fibromyalgia (FM) is a chronic disorder marked by widespread musculoskeletal pain, fatigue, sleep disturbances, and cognitive difficulties. Patients often experience hyperalgesia, allodynia, and muscle weakness. Central sensitization plays a key role, making the nervous system more responsive to pain. Though muscles are mainly affected, joint pain, stiffness, and reduced mobility are also common. Chronic pain and poor posture can worsen musculoskeletal health. FM is not mainly inflammatory, but pain and stress may affect bone health. Sleep disorders, like non-restorative sleep and apnea, are frequent and worsen fatigue. Neurotransmitter imbalances (e.g., serotonin, dopamine) affect pain and muscle function.

The American College of Rheumatology defines FM by widespread bilateral pain lasting at least three months. FM mainly affects women, with a prevalence of 0.2-6.6%, often starting between the ages of 30 and 35. Besides physical symptoms, many patients suffer from anxiety, depression, and mood disorders, affecting their quality of life.

Gastrointestinal issues, especially irritable bowel syndrome (IBS), are also frequent in FM patients. Both conditions share mechanisms such as pain hypersensitivity, altered autonomic regulation, gut-brain axis disruption, and immune dysfunction. Low-grade inflammation and intestinal permeability may contribute to chronic symptoms.

FM treatment includes anticonvulsants, antidepressants, and painkillers. IBS is managed with diet changes and medications like antispasmodics. Due to limited drug effectiveness, multidisciplinary approaches are gaining attention. Physical exercise is a proven non-drug strategy that improves pain, fatigue, and mental health in FM and IBS. Still, adherence is low due to fear of pain, fatigue, and low motivation.

Exercise, especially aerobic activity, benefits IBS patients by improving gut symptoms and reducing inflammation. It may also strengthen the gut barrier in both conditions. While optimal programs need more study, exercise is a promising therapy. Major health bodies recommend aerobic, resistance, and flexibility training for FM and aerobic exercise for IBS.

DETAILED DESCRIPTION:
Patient Recruitment: The study is designed as a randomized crossover trial. Patients will be recruited from the "Rheumatology," "Pain Therapy," and "Celiac Disease and Functional Disorders" adult (30-65 years) outpatient clinics at the IRCCS "S. de Bellis" in Castellana Grotte (BA). Recruitment will take place following the confirmation of a diagnosis of irritable bowel syndrome (IBS) concomitant with fibromyalgia (FM).

Information regarding the participant's health status will be gathered through a comprehensive visit, encompassing an interview covering lifestyle, medical history, and a physical examination. Additionally, metabolic parameters, including blood sugar, HbA1c, lipid profile, and body weight, must fall within the normal range of values. Before providing written consent, all participants will receive verbal and written details of the study. The recruitment and evaluation of patients will be structured into the following phases:

V0. The patients will receive information about the study, sign an informed consent form, and complete a clinical history form. They will also maintain a daily symptom diary for 14 days. Furthermore, after confirming the inclusion criteria, participants will receive an accelerometer for 7 days to monitor their physical activity levels and sleep quality.

V1. Subjects will undergo blood sampling, urine, and stool sample collection, completion of questionnaires on gastrointestinal (GI) symptoms, fibromyalgia (FM), psychology, quality of life (QoL), and physical activity, as well as anthropometric measurements and bioimpedance analysis. Before the physical exercise intervention, field tests for physical fitness will be conducted, including handgrip strength tests, walking tests, and flexibility assessments. After obtaining certification of physical fitness for non-competitive sports activities, patients will be instructed to participate in a specific exercise program under the supervision of exercise specialists.

V2. Patients will repeat the GI, FM, psychology, QoL, and physical activity questionnaires. They will undergo the same functional tests and report adverse events. Blood and biological samples will be collected, and accelerometers will be worn for 7 days to assess changes in physical activity and sleep quality.

Washout Period. The washout period will last 4 weeks, during which recruited subjects will be returned as closely as possible to their baseline conditions. After these 60 days, subjects will be recalled, undergo the same evaluations, and be invited to participate in various physical exercise programs.

V3. During this visit, all evaluations from V1 will be repeated. Patients will also be asked to wear the accelerometer for seven days.

V4. During this visit, all evaluations from V2 will be repeated. All examinations will take place at the IRCCS "S. de Bellis," while motor tests and training sessions will be conducted at a gym affiliated with the institute.

Evaluation of FM Symptoms: To assess FM symptoms, a series of validated questionnaires, some specific to FM and others more general (e.g., the Fibromyalgia Impact Questionnaire, modified version (FIQ-R), Digital Tender Point examination, Brief Pain Inventory (BPI), and Pittsburgh Sleep Quality Index (PSQI) ), are utilized.

Evaluation of GI Symptoms: A patient's clinical history form is completed before assessing GI symptoms. Subsequently, two questionnaires are administered: the IBS-SSS, specific to IBS symptoms.

Psychological Assessment: The psychological profile is assessed using validated questionnaires. Initially, a history form identifies prior psychopathological disorders or family history. Additionally, first and second-level stress factors linked to symptoms are pinpointed. At baseline and day 120, participants complete pre- and post-administered psychological questionnaires covering various aspects, including the Symptom Checklist (SCL)-90-R, Perceived Stress Scale (PSS), World Health Organization Quality of Life-Brief (WHOQOL-Brief), Delaying Gratification Inventory (DGI), Rotter's Locus of Control Scale, Subjective Happiness Scale (SHS), Attachment Style Questionnaire (ASQ), and Psychological Well-Being Scales (PWBS).

Anthropometric and Bioimpedance Assessment: The subjects' physical characteristics (body weight, height, and circumferences) are assessed through direct measurement. Bioimpedance measurement involves a non-invasive, rapid, and quickly executed examination, ideal for measuring nutritional status (lean mass, fat mass, cellular and muscle mass), hydration status (water retention, swelling, hyperhydration, inflammation), basal metabolism, and "ideal weight".

Evaluation of Intestinal Permeability (IP): IP will be evaluated at baseline (day 0) and day 120. This involves administering a mixture of 40 g sucrose, 10 g lactulose, 5 g mannitol, and 1 g sucralose and measuring their gastrointestinal (GI) absorption through urinary excretion of these sugars. Urine will be collected over the next 5 hours in containers with added chlorhexidine (500 µL) as a preservative. The different sugars in the urine will be determined using high-pressure liquid chromatography (HPLC) and subsequent pulsed amperometric detection. Results will be expressed as a percentage of the excreted sugars in urine relative to the administered amount.

Barrier Peptide Assay: Zonulin, intestinal fatty acid binding protein (I-FABP), diamine oxidase (DAO), and D-lactate assays will be conducted at baseline (day 0) and day 120 using commercially available Enzyme-Linked Immunosorbent Assay (ELISA) methods.

Indole and Skatole Assay: Indole will be assayed using a colorimetric analytical method, while skatole will be assessed using a refined chromatographic method with fluorimetric detection. Both assays will be conducted on a urine sample. This investigation will be conducted at baseline and day 120.

Biochemical analyses: blood levels of interleukin (IL)-6, IL-8, IL-10, tumor necrosis factor (TNF)-alpha, and peptides involved in the regulation of GI motility (somatostatin, motilin, serotonin, somatostatin, motilin, serotonin, etc.)

Physical Activity Assessment: Physical activity levels will be measured using the International Physical Activity Questionnaire (IPAQ short-form) and accelerometer (ActiGraph GT9X Link), which will monitor physical activity and sleep quality. Additionally, participants will complete the Tampa Scale of Kinesiophobia (TSK) to assess their fear of movement.

Field tests will be conducted to evaluate physical fitness, including the 2 km walk test, Six Minutes Walking Test, Hand Grip Test, Sit and Reach Test, 30'' Sit to Stand test, Step Test, and Single Leg Stance (SLS). During the tests, symptoms, pain severity, fatigue, and exercise experience will be monitored in patients with fibromyalgia. Participants will be informed about the differences between exercise-induced soreness and pain/fatigue associated with fibromyalgia.

Treatments

Subjects will be randomized into two different intervention groups:

Treatment 1: A specific nutritional plan for individuals with IBS combined with a combined exercise program (CE).

Treatment 2: A specific nutritional plan for individuals with IBS combined with an aerobic exercise program (AE).

Intervention Protocol Based on existing literature, two interventions have been selected to identify the optimal exercise protocol for managing FM and IBS. The American College of Sports Medicine (ACSM) recommends combined exercise for FM, while aerobic exercise is effective for IBS. This study compares the two protocols to determine which is more suitable for individuals with both conditions, aiming to identify the most effective therapeutic approach.

Combined Exercise (CE) Frequency: 3 times per week for 4 months, on non-consecutive days. Intensity: Monitored with a heart rate monitor and personalized using Tanaka's formula. Additionally, the TALK TEST (a standardized, validated tool based on the subject's ability to maintain a conversation during exercise) and the Borg Scale will be used to measure exertion.

Aerobic Activity: 60-75% of max heart rate. Resistance: 6/7 on the Borg Scale. Flexibility: Range of motion (ROM) without pain. Type: Moderate aerobic exercise combined with resistance and flexibility exercises.

Aerobic Activity: Low-impact, non-weight-bearing exercises to minimize exercise-induced pain.

Resistance Activity: Circuit training with small equipment (resistance bands, dumbbells, ankle or wrist weights).

Flexibility Exercises: Stretching with and without bands. Duration: 60-minute sessions, including warm-up, aerobic, strength, and flexibility exercises, and cool-down, twice a week.

One specific session per week will focus on flexibility exercises. Joint mobility and flexibility exercises will be performed dynamically and statically after 20 minutes of aerobic exercise on machines.

Aerobic Exercise (AE) Frequency: 3 times per week for 4 months, on non-consecutive days. Intensity: Monitored with heart rate monitor, Tanaka's formula, TALK TEST, and Borg Scale. Aerobic activity at 60-75% of max heart rate.

Type: Low-impact, non-weight-bearing aerobic exercise. Duration: 60-minute sessions, including warm-up, aerobic activity, small circuits, and cool-down.

Both intervention protocols will be performed in small groups under the supervision of graduates in preventive and adapted exercise science. The exercise volume will be adjusted accordingly if symptoms worsen during group activities. Intensity or duration will be reduced before frequency to maintain regular activity.

Primary Endpoint: Perceived physical function will be assessed using the total score of the FIQ-R (higher scores indicate poorer functioning). The expected outcome is a 20% improvement in the total FIQ-R and IBS-SSS scores at the end of the intervention.

Secondary Endpoints: The effects of physical exercise on physical efficacy, dysbiosis, systemic inflammation, microbiota, and psychological profile will also be investigated.

Statistical Analysis:

Data will be presented as mean (SD) or median and 5th and 95th percentiles, depending on whether the variables are continuous or categorical. All comparisons will be made using non-parametric tests to avoid assuming a normal data distribution. Proportions related to dichotomous variables will be compared using the Chi-square test. P-values <0.05 (two-tailed) will be considered statistically significant. All patients receiving physical activity instructions will be included in the statistical analysis for data comparison at the end of the treatment period, with dropouts categorized as non-responders (Intention To Treat analysis). The comparison of post-intervention data versus baseline will be conducted only for those who completed the intervention (per-protocol analysis). All statistical analyses will be performed using SigmaSTAT (Systat Software, Inc., San Jose, CA, USA) and GraphPad Prism 5 (GraphPad Software Inc., La Jolla, CA, USA). Questionnaire data will be entered into a database by a person not involved in the study.

Study Power Calculation:

The sample size is calculated to detect a 39% improvement in the total IBS-SSS score before and after the intervention. Considering a standard deviation of 30, a power of 0.80, and a significance level of 0.05, a minimum of 11 patients per group must be recruited. With a 27% dropout rate, each group will comprise 15 patients (total = 30).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Irritable Bowel Syndrome (IBS) concomitant with Fibromyalgia (FM).Meeting the American College of Rheumatology (ACR) diagnostic criteria for FM and meeting the Rome III/IV diagnostic criteria for IBS.
* Total score on the Irritable Bowel Syndrome Severity Scoring System (IBS-SSS) ≥ 125 (indicating moderate to severe IBS symptoms).
* Men and women aged between 30 and 65 years.
* Body Mass Index (BMI) between 18.5 and 29.9.

Exclusion Criteria:

* Individuals with severe cardiac, hepatic, neurological, psychiatric disorders, or other gastrointestinal diseases.
* Individuals unable to discontinue symptom management therapies and medications for FM/IBS.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Fibromyalgia symptom assesment | At baseline and day 120
  To evaluate the effectiveness of an exercise intervention on IBS symptoms as measured by a change in the Fibromyalgia Impact Questionnaire, modified version (FIQ-R) scores from baseline.
  The FIQ serves as a tool for assessing and evaluating the condition of patients with fibromyalgia (FM) and tracking their progress and outcomes. Specifically designed to gauge the aspects of health status most impacted by FM, the FIQ comprises ten items. The initial item consists of 11 questions about physical functioning, each rated on a 4-point Likert-type scale. The subsequent items (2 and 3) prompt patients to indicate the number of days they felt well and the days they were unable to engage in work or housework due to FM symptoms. Items 4 through 10 feature horizontal linear scales with ten increments, allowing patients to rate work difficulty, pain, fatigue, morning tiredness, stiffness, anxiety, and depression.
IBS symptoms assessment | At baseline and day 120
  To evaluate the effectiveness of an exercise intervention on IBS symptoms as measured by a change in the IBS-Symptom Severity Scale (IBS-SSS) questionnaire score from baseline.
  The IBS-SSS is a validated questionnaire for gastrointestinal symptoms and provides a global measure of symptom severity by assessing five items ("severity of abdominal pain", "frequency of abdominal pain", "severity of abdominal distension", "dissatisfaction with bowel habits", "impact of symptoms on quality of life") on a visual analog scale. The values of the five items are added together to give a total score between 0 and 500. Cases are then classified as 'mild' (75 to 175), 'moderate' (175 to 300) and 'severe' (>300).

SECONDARY OUTCOMES:
Physical Fitness assessment | Al Baseline and day 120
  Field tests to assess participants' physical fitness include the 2 km Walk Test, which evaluates cardiovascular fitness by recording heart rate and walking time before and after the test. The Six-Minute Walk Test measures aerobic fitness and functional capacity, requiring participants to walk as far as possible in 6 minutes, with heart rate monitored and exertion assessed using the Borg Scale. The Hand Grip Test assesses maximum hand and forearm strength using a dynamometer, with three tests per hand and the average recorded. The Sit and Reach Test measures flexibility in the back and legs, recording the best of two attempts. The 30-second Sit to Stand Test evaluates lower limb strength and endurance by counting the number of complete sit-to-stand movements in 30 seconds without using arms for support. The Step Test assesses cardiovascular endurance and lower limb function by having participants repeatedly step onto a standard-height step for 3 minutes, with recovery heart rate record
Psychological Assessment: | At baseline and day 120
  The Symptom Checklist (SCL)-90-R questionnaire will evaluate the psychological profile
  The Symptom Checklist-90-Revised (SCL-90-R) is a widely employed self-report questionnaire in clinical and research settings. It aims to evaluate diverse psychological symptoms and distress in individuals. Comprising 90 items, the SCL-90-R addresses dimensions of psychological well-being and psychopathology, including somatization, obsessive-compulsive symptoms, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, and psychoticism. Respondents use a Likert scale ranging from 0 (not at all) to 4 (extremely) to rate the extent of their experience with each symptom over a specified timeframe, typically the past week. This questionnaire offers a comprehensive profile of an individual's psychological symptoms, aiding in identifying areas of distress or dysfunction.
Evaluation of Barrier Peptide Integrity | At baseline and day 120
  Zonulin, I-FABP, DAO, and D-lactate assays will be performed using commercially available ELISA assays for each peptide.
Intestinal microbiota analysis | At baseline and day 120
  Any differences in the intestinal microbial population in the different disease patterns considered will be evaluated using appropriate genetic and molecular investigations (Illumina/Solexa Genetic Analyzer HiSeq) on the patient's stool samples.
Evaluation of Intestinal dysbiosis | At baseline and day 120
  The intestinal dysbiosis will be evaluated by assaying Indole using a colorimetric analytical method as a marker of fermentative dysbiosis, Skatole, a marker of putrefactive dysbiosis, will be assessed using a refined chromatographic method with fluorimetric detection. Both assays will be conducted on a urine sample.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Saverio de Bellis, Castellana Grotte, Bari, Italy